CLINICAL TRIAL: NCT02745106
Title: Randomized Pilot Trial of Interventional Treatment of Residual Pulmonary Hypertension in Patients After Pulmonary Thromboendarterectomy
Brief Title: Interventional Treatment of Residual Pulmonary Hypertension in Patients After Pulmonary Thromboendarterectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Novosibirsk Scientific Research Institute for Circulatory Pathology (Other)
Responsible Party: Principal Investigator, Alexander Edemskiy, Principal investigator Alexander Edemskiy, Novosibirsk Scientific Research Institute for Circulatory Pathology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PADN1
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic thromboembolic pulmonary hypertension, Navigation system, Ablation
MeSH Terms: interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PADN treatment (Experimental): Procedure/Surgery: Right heart catheterization, Radiofrequency pulmonary artery denervation using following devices:
  1. Ablation catheter
  2. Carto 3, Carto RMT, Stereotaxis
  3. Swan-Ganz catheter
  Interventions: Procedure: Radiofrequency pulmonary artery denervation; Device: Ablation catheter; Device: Swan-Ganz catheter for right heart catheterization
- Control (Sham) (Sham Comparator): Procedure: Right heart catheterization
  Using following device:
  - Swan-Ganz catheter
  Interventions: Device: Swan-Ganz catheter for right heart catheterization

INTERVENTIONS:
Procedure: Radiofrequency pulmonary artery denervation — Radiofrequency ablation of pulmonary artery will be performed with standard electrophysiological catheter and non-fluoroscopic 3D-navigation system. Right heart catheterization (thermodilution method with Swan-Ganz catheter) will be performed before and after procedure. The radiofrequent impact will be performed 2mm after pulmonary artery bifurcation in both right and left main pulmonary artery branches. The radiofrequent impact will be performed at temperature 40-42 C, up to 12 watts and 60 second duration in every ablation point under impedance control.
  Other Names: PADN
  Arms: PADN treatment
Device: Ablation catheter — 4MM RF CONDUCTR (MULTI-CURVE) SERIES ABLATION CATHETER Standart procedure for radiofrequency ablation: Radiofrequency ablation of pulmonary artery will be performed with standard electrophysiological catheter and non-fluoroscopic 3D-navigation system. Right heart catheterization (thermodilution method with Swan-Ganz catheter) will be performed before and after procedure. The radiofrequent impact will be performed 2mm after pulmonary artery bifurcation in both right and left main pulmonary artery branches. The radiofrequent impact will be performed at temperature 40-42 C, up to 12 watts and 60 second duration in every ablation point under impedance control.
  Arms: PADN treatment
Device: Swan-Ganz catheter for right heart catheterization — Standart procedure of right catheterization:
  * punction of right jugular vein with Seldinger technique, introducer placement
  * insertion of Swan-Ganz catheter via introducer in jugular vein under fluoroscopic control and wave form of monitor's curve.
  * positioning of swan-ganz catheter in pulmonary artery
  * direct central hemodynamics measurements: systolic/diastolic/mean pulmonary artery pressure, pulmonary capillary wedge pressure, cardiac output (thermodilution technique)
  * calculating of indirect parameters (pulmonary vascular resistance)

SUMMARY:
The study evaluates the technique of non-drug treatment of residual pulmonary hypertension in patients with chronic thromboembolic pulmonary hypertension after pulmonary thromboendarterectomy.

DETAILED DESCRIPTION:
The best strategy of treatment patients with chronic thromboembolic pulmonary hypertension is pulmonary thromboendarterectomy. In 5-30% of cases after pulmonary thromboendarterectomy residual pulmonary hypertension is persisted. The technique of radiofrequency pulmonary artery denervation in patients with idiopathic pulmonary arterial hypertension (type I) is known and was assessed during clinical investigation. In this study radiofrequency pulmonary artery denervation technique may be applied in patients with residual pulmonary hypertension after pulmonary thromboendarterectomy (type IV)

ELIGIBILITY:
Inclusion Criteria:

* presence of residual pulmonary hypertension in patients after pulmonary thromboendarterectomy according to right heart catheterization: mean pulmonary artery pressure > 25 mm Hg or pulmonary vascular resistance > 400 dyn x sec x cm-5

Exclusion Criteria:

* no evidence of residual pulmonary hypertension in patients after pulmonary thromboendarterectomy (mean pulmonary artery pressure <25 m Hg).
* refusal of a patient to participate in the study.
* the presence of severe concomitant diseases of the cardiovascular system and lungs, leading to pulmonary hypertension
* the presence of other severe comorbidities that may result in death within a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance | 12 months
  Units - (dyn x sec x cm-5)

SECONDARY OUTCOMES:
6-minute walking distance test | 12 months
Echocardiographical sings of right ventricle function - 1 | 12 months
  Fractional area change (%)
Echocardiographical sings of right ventricle function - 2 | 12 months
  Tricuspid annular systolic excursion, TAPSE (mm)
Pulmonary artery pressure | 12 months
  Pulmonary artery pressure (systolic/diastolic/mean) will be measured by right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chernyavskiy, PhD, Study Chair — 15 Rechkunovskaya street, Novosibirsk, Russia, 630055; Alexander Romanov, PhD, Study Chair — Novosibirsk Scientific Research Institute for Circulatory Pathology; Evgeny Pokushalov, PhD, Study Chair — Novosibirsk Scientific Research Institute for Circulatory Pathology
Locations (1):
- Novosibirsk research institute of circulation pathology, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes